CLINICAL TRIAL: NCT00160277
Title: Open Label, Multi-Center, Force-Titration Study to Evaluate the Efficacy and Safety of Moxonidine in Ambulatory Subjects With Essential Hypertension
Brief Title: Efficacy and Safety of Moxonidine in Indian Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S220.3.124
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension
Keywords: Efficacy and safety of moxonidine in Indian hypertensives
MeSH Terms: conditions — Hypertension | interventions — moxonidine

INTERVENTIONS:
Drug: Moxonidine

SUMMARY:
The purpose of this study is to demonstrate efficacy and safety of Moxonidine in Indian subjects.

ELIGIBILITY:
Inclusion Criteria:

Hypertension

Exclusion Criteria:

Severe concomitant diseases, CHF, secondary hypertension, severe hypertension, significant hepatic disease, unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07

PRIMARY OUTCOMES:
Systolic blood pressure reduction

SECONDARY OUTCOMES:
Piggy-back pharmacoeconomic evaluation; Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- India (3):
  - Site 1, Jubillee Hills Hyderabad
  - Site 2, Mangalore
  - Site 3, New Delhi